CLINICAL TRIAL: NCT04127175
Title: Breast Density Measurements in Digital Mammography and Breast Tomosynthesis Systems of Different Pixel Size
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: University of Barcelona (Other); Universitat de Girona (Other)
Responsible Party: Principal Investigator, Oliver Diaz-Montesdeoca, Visiting researcher, Corporacion Parc Tauli
Other Study IDs: 2019/629
Record Dates: First submitted 2019-10-12; First posted 2019-10-15 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Mammographic Breast Density
Keywords: Breast cancer; Breast density; Volpara; Quantra; BI-RADS; Digital Mammography; Digital Breast Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Volpara — This tool represents a physics-based model which extract pixel-wise information from the FFDM or DBT images, and combine it with metadata information from the DICOM header and appropriate linear attenuation coefficients of both adipose and glandular tissue.

SUMMARY:
Breast cancer (BC) is the most frequently diagnosed cancer in women worldwide. The cause of developing BC is currently unknown. However, there are several risk factors, such as volumetric breast density (VBD), which have been proved to have a relationship with BC. The assessment of breast density is typically performed subjectively using the 4-classes density classification described by American College of Radiology. However, in the last years, automated breast density software tools have been developed (e.g. Volpara, Quantra). In this work, VBD measurements from VolparaTM (v. 1.5.4.0) will be compared between Full-Field Digital Mammography (FFDM) and Digital Breast Tomosynthesis (DBT) of the same pacient ('combo mode'). Images will be acquired in a Hologic Selenia Dimensions, the most common FFDM/DTB system, where image resolution is different for FFDM (70 um) and DBT (140 um).

This study (1) evaluates the consistency between Volpara's breast density measurements and spatial distribution for the two imaging techniques (FFDM and DBT) in a Hologic Selenia Dimensions, and (2) compares VDB measurements with other similar tool (Quantra) and radiologists breast density manual classification.

DETAILED DESCRIPTION:
Monocentric, prospective and observational study which will analyse a series of 300 cases (FFDM + DBT) from consecutive women. Image acquisitions will take place within the Área de radiología Mamaria y Ginecológica located at Parc Taulí Hospital Universitari, Sabadell. The purposes of this study will be explained to each potential candidate and if agreed to participate, a consent form will be signed.

Inclusion criteria:

* Subjects over 18 years old.
* Acceptance of participation through a signed consent form.
* Asymptomatic subjects

Exclusion criteria:

* Subjects refusing to participate or sign the consent form.
* Subjects with prior history of breast surgery or biopsy with markers.
* Subjects with breast prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of participation through a signed consent form.
* Asymptomatic subjects

Exclusion Criteria:

* Subjects refusing to participate or sign the consent form.
* Subjects with prior history of breast surgery or biopsy with markers.
* Subjects with breast prostheses.
* Subjects with biopsy marker clips

Ages: 40 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Asymptomatic women with age greater than 40 who has signed a consent form.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Consistency of breast density measurements from the latest VolparaTM breast density tool for Hologic's FFDM and DBT images (i.e. combo mode). | 1 year
Comparison of VolparaTM's Volumetric Breast Density measurements and its 4-classes density rating measured in DBT against QuantraTM 3D and radiologist's BI-RADS manual classification | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology Breast Unit, Hospital Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Breast density software which will be evaluated — https://volparasolutions.com/science-hub/breast-density/measuring-breast-density